CLINICAL TRIAL: NCT04900974
Title: Single Dose Pharmacokinetics of Doravirine in HIV-infected Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0052
Record Dates: First submitted 2021-05-13; First posted 2021-05-25 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Pregnancy Related
MeSH Terms: conditions — HIV Infections | interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doravirine (Experimental): 100mg doravirine given by mouth once at each sampling visit.
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — 100mg

SUMMARY:
The purpose of this research study is to evaluate the effect of body changes in pregnancy on doravirine concentrations, to determine what dose of doravirine should be used. Study participants will remain on their normal antiretroviral medications (ARVs) while participating in this study as prescribed by their regular clinic provider. Study participants will come to the research clinic for three sampling visits throughout their time as a participant. Study participants will only take one dose of doravirine during each sampling visit, which will occur during the 2nd and 3rd trimesters, as well as after their baby is delivered. This study was designed intentionally to not give a dose of doravirine in the first trimester when there is the greatest chance for all drugs to potentially cause injury to the baby. Study participants that choose to participate in this study may be enrolled for up to 10 months depending on the length of their pregnancy and how the visits are scheduled.

DETAILED DESCRIPTION:
Antiretroviral (ARV) medications are used to treat infection with human immunodeficiency virus (HIV). During pregnancy, ARV therapy keeps women healthy and decreases the spread of HIV to their babies (<1-2%).

Many changes occur in the body during pregnancy, which can alter the concentrations of drug in the body. Doravirine (DOR) is a Food and Drug Administration (FDA) approved ARV, but the extent to which the drug concentrations of doravirine change during pregnancy is unknown. Because these changes are unknown, DOR has not been approved by the FDA for use among pregnant women; however, the FDA has given the researchers permission to use it in this study Pregnant women are often excluded from clinical trials, so it can take several years after a drug gets approved before contemporary ARV is available to them.

The purpose of this research study is to evaluate the effect of body changes in pregnancy on doravirine concentrations, to determine what dose of doravirine should be used. Study participants will remain on their normal antiretroviral medications (ARVs) while participating in this study as prescribed by their regular clinic provider. Study participants will come to the research clinic for three sampling visits throughout their time as a participant. Study participants will only take one dose of doravirine during each sampling visit, which will occur during the 2nd and 3rd trimesters, as well as after their baby is delivered. This study was designed intentionally to not give a dose of doravirine in the first trimester when there is the greatest chance for all drugs to potentially cause injury to the baby. Study participants that choose to participate in this study may be enrolled for up to 10 months depending on the length of their pregnancy and how the visits are scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women living with Human Immunodeficiency Virus (HIV) ≥18 years of age
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the trial.
* On stable combination Antiretroviral Therapy (cART) for at least 30 days prior to enrollment
* Plasma HIV RNA < 50 copies/mL within 90 days prior to enrollment
* Ability and willingness of participant to not change their cART regimen to avoid any confounding of pharmacokinetic (PK) parameters.

  o Note: Women who change cART regimens will be replaced.
* Aspartate aminotransferase and alanine aminotransferase < 3x Upper Limit of Normal (ULN)
* Hemoglobin lower than Division of AIDs (Acquired Immunodeficiency Syndrome) (DAIDs) Grade 2 (9.0 g/dL)

Exclusion Criteria:

* Women with multiple gestation, active opportunistic infections, present obstetrical complications that would deem them unsuitable for study participation, or evidence of fetal anomalies in present pregnancy will be excluded.
* Women with severe renal impairment, end stage renal disease, undergoing dialysis, or severe hepatic impairment (Child-Pugh C)
* Women with a significant illness/condition at the time of enrollment that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or assessment of safety.
* Women with pregnancies that have become complicated are excluded for safety reasons.
* Active hepatitis C (HCV) infection as defined by anti-hepatitis C virus serology (as determined by multi-antigen EIA) and detectable HCV RNA.
* Clinically significant labs greater than Grade 2 on the NIH Division of AIDs Table for Grading the Severity of Adult and Pediatric Adverse events
* Receiving CYP3A inducers including carbamazepine, phenobarbital, phenytoin, enzalutamide, rifampin, rifapentine, mitotane, or St. John's wort or other drugs, including antiretrovirals, that influence drug concentration or alter pharmacokinetic profiles (atazanavir, maraviroc, darunavir, norvir, efavirenz, tipranavir)
* Receiving moderate to strong cytochrome p450 3A (CYP3A) inhibitors including clarithromycin, boceprevir, cobicistat, danoprevir and ritonavir, elvitegravir and ritonavir, indinavir and ritonavir, itraconazole, ketoconazole, lopinavir and ritonavir, paritaprevir and ritonavir, posaconazole, ritonavir, saquinavir and ritonavir, telaprevir, tipranavir and ritonavir, grapefruit juice, idelalisib, nefazodone, and nelfinavir.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Change in total and protein-unbound Cmax of doravirine in blood plasma during pregnancy. | Pre-dose (within 1 hour prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 and hours post-dose in each period.
  To describe single-dose total and protein-unbound Cmax of doravirine in the blood plasma of women living with HIV during the 2nd trimester, 3rd trimester, and post-partum
Change in total and protein-unbound Tmax of doravirine in blood plasma during pregnancy. | Pre-dose (within 1 hour prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 and hours post-dose in each period.
  To describe single-dose total and protein-unbound Tmax of doravirine in the blood plasma of women living with HIV during the 2nd trimester, 3rd trimester, and post-partum
Change in total and protein-unbound C12h of doravirine in blood plasma during pregnancy. | Pre-dose (within 1 hour prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 and hours post-dose in each period.
  To describe single-dose total and protein-unbound C12h of doravirine in the blood plasma of women living with HIV during the 2nd trimester, 3rd trimester, and post-partum
Change in total and protein-unbound C24h of doravirine in blood plasma during pregnancy. | Pre-dose (within 1 hour prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 and hours post-dose in each period.
  To describe single-dose total and protein-unbound C24h of doravirine in the blood plasma of women living with HIV during the 2nd trimester, 3rd trimester, and post-partum
Change in total and protein-unbound Area Under the Curve (AUC) of doravirine in blood plasma during pregnancy. | Pre-dose (within 1 hour prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 and hours post-dose in each period.
  To describe single-dose total and protein-unbound AUC of doravirine in the blood plasma of women living with HIV during the 2nd trimester, 3rd trimester, and post-partum

SECONDARY OUTCOMES:
Number of Adverse Events reported after single doses of doravirine in pregnant participants. | From enrollment visit to follow-up visit, an average of 10 months.
  To evaluate the number of Adverse Events reported after single doses of doravirine in pregnant participants living with HIV

CONTACTS AND LOCATIONS:
Overall Officials: Angela Kashuba, PharmD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 9 to 36 months following publication.